CLINICAL TRIAL: NCT05875389
Title: Virtual Intervention Stroke Initiative by Ottawa Neurology
Brief Title: Virtual Intervention Stroke Initiative
Acronym: VISION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230211-01H
Record Dates: First submitted 2023-05-09; First posted 2023-05-25 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Stroke; Acute Ischemic Stroke
Keywords: telemedicine; virtual care
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual assessment (Experimental): virtual assessment with a stroke neurologist/advanced practice nurse, with interdisciplinary support, to facilitate the care of patients admitted to primary stroke centres using existing tools for remote evaluation and review.
  Interventions: Other: Virtual assessment

INTERVENTIONS:
Other: Virtual assessment — virtual assessment with a stroke neurologist/advanced practice nurse, with interdisciplinary support, to facilitate the care of patients admitted to primary stroke centres using existing tools for remote evaluation and review.

SUMMARY:
The goal of this clinical trial is to determine if patients admitted to a primary stroke centre, such as the general internal medicine service of the Ottawa Hospitals General Campus, for acute ischemic stroke would benefit from a scheduled virtual assessment with a stroke neurologist to review investigations, results, and evaluations to identify stroke etiology, propose appropriate therapy, and guide decision-making and multidisciplinary assessment, similar to services provided to patients admitted to comprehensive stroke centres, such as the Civic Campus of the Ottawa Hospital.

DETAILED DESCRIPTION:
Patients admitted to primary stroke centres do not have access to the same level of stroke expertise on site as do patients admitted to comprehensive stroke centres, resulting in increased length of stay with implications for access to stroke rehabilitation. Virtual access to stroke experts has been used in hyperacute stroke care through programs such as Ontario Telestroke, but this has not been routinely used for acute inpatient management. The investigators propose a system to provide virtual access to the stroke neurology team to patients admitted with stroke in a primary stroke centre. Patients at the General Campus of the Ottawa Hospital are currently admitted to Internal Medicine; this includes scheduled virtual assessment with a stroke neurologist and advanced practice nurse/interdisciplinary support to review investigations, results, and evaluations to identify stroke etiology, propose appropriate therapy, and guide decision-making and multidisciplinary assessment, similar to services provided to patients admitted to the Civic Campus. This will be developed with the assistance of Internal Medicine and will utilize technologies and assessment tools and strategies already being used for provision of virtual care in other settings. The goal of this project will be to prove that patients in primary stroke centres, with the assistance of virtual care, can benefit from the expertise available at comprehensive centers throughout their stay, and that this will result in an improved quality of care with benefits for patients, hospitals, and the community.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* admitted to the general internal medicine service of the Ottawa Hospital General Campus for acute ischemic stroke
* able to participate in video assessments with necessary accommodation/facilitation for participation (particularly if stroke results in physical or communication deficits)

Exclusion Criteria:

* patients who are unable, in the judgement of the study team or treating team, to participate in video assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Morbidity-adjusted length of stay | Through study completion, an average of 6 months
  Number of days admitted to general internal medicine

SECONDARY OUTCOMES:
Length of time on ALC | Through study completion, an average of 6 months
  Length of time on alternate level of care

OTHER OUTCOMES:
Discharge destination | Over 6 months
  The classification of where a patient is sent on completion of their hospital admission (i.e. home vs. rehabilitation vs. other facility vs. death)
Functional outcome | Over 6 months
  modified Rankin Score 0-6 (0 is no symptoms at all, and 6 is death)
Home time | Over 6 months
  patient-centered metric examining time spent at home after discharge from hospital/rehabilitation at 6 months

IPD SHARING:
Plan to Share IPD: No